CLINICAL TRIAL: NCT07171151
Title: Measurement of MMP-8, MMP-9, RANKL, MIP-1alpha in Biopsy Samples From Odontogenic Cyst Patients
Brief Title: Detection of Disease Marker Factors in Cyst Fluid
Status: Recruiting | Type: Observational
Sponsor: Harran University (Other)
Responsible Party: Principal Investigator, mine alkaya karagoz, Assistant Professor, Harran University
Other Study IDs: HRU/25.11.54
Record Dates: First submitted 2025-08-25; First posted 2025-09-12 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Biomarkers
Keywords: odontogenic cysts; biomarkers; MMP-8; MIP-1alfa
MeSH Terms: conditions — Odontogenic Cysts

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Weeks
Biospecimen Retention: Samples With DNA — Cyst fluid obtained during puncture
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- individuals with odontogenic cysts: The cyst fluid obtained during the puncture will be collected in a tube and centrifuged. The clear liquid remaining on top will be transferred to an Eppendorf tube and stored at -80 degrees. After all samples are collected, they will be analyzed using the ELISA method.
  Interventions: Other: cyst fluid examination

INTERVENTIONS:
Other: cyst fluid examination — Participants will not undergo any procedures outside of the routine for the study. The cyst fluid obtained during the puncture will be collected in a tube and centrifuged at 3000 rpm for 20 minutes at 4 degrees Celsius. The Eppendorf tubes will be stored at -80 °C until the clear liquid remaining above is taken and examined, without removing the particles that have settled at the bottom of the tube. The biochemical parameters of the cyst fluid obtained from the study participants will be analyzed using the ELISA method. MMP-8, MMP-9, RANKL, and MIP1alpha will be analyzed using commercially available ELISA kits, following the manufacturer's instructions.

SUMMARY:
The purpose of this observational study is to examine the cyst fluid obtained after a puncture procedure performed for cyst diagnosis in participants with cystic lesions on clinical and radiological examination.The main question it aims to answer is:

- What is the exact mechanism of formation of odontogenic cysts?

Biomarkers in the cyst fluid obtained after a puncture procedure performed as part of the diagnosis and treatment process of odontogenic cysts will be examined. The aim of this study is to gain insight into cyst pathology by examining the levels of biomarkers in odontogenic cyst fluid.

DETAILED DESCRIPTION:
Patients with cystic lesions who apply to Harran University Oral and Maxillofacial Surgery between August 2025 and December 2025 will be included in the study. Approximately 25 patients are planned to be included in the study. Informed consent will be obtained from patients included in the study.

Participants will not undergo any procedures outside of the routine for the study. Aspiration will be performed before cyst enucleation/marsupialization. Later, excisional/incisional biopsies will also be performed during enucleation and marsupialization.The cyst fluid obtained during the puncture will be collected in a tube and centrifuged at 3000 rpm for 20 minutes at 4 degrees Celsius. The Eppendorf tubes will be stored at -80 °C until the clear liquid remaining above is taken and examined, without removing the particles that have settled at the bottom of the tube. The biochemical parameters of the cyst fluid obtained from the study participants will be analyzed using the ELISA method. MMP-8, MMP-9, RANKL, and MIP1alpha will be analyzed using commercially available ELISA kits, following the manufacturer's instructions.

While the concentration levels of MMP-8, MMP-9, RANKL, and MIP-1alpha are dependent variables, the cyst type, its inflammatory or developmental origin, and other clinical features are independent variables.The data will be calculated using the SPSS program. The normality of the data will be examined using the Shapiro-Wilk and Kolmogorov tests, and outliers will be calculated using boxplots and Z-scores. When comparing variables with a normal distribution in two independent groups, the "independent samples t-test" will be used; if there is no normal distribution, the Mann-Whitney U test will be used. If three or more distributions are normal, "one-way ANOVA" will be used; if normal distribution is not found, the Kruskal-Wallis test will be used. If the data is normally distributed, the Pearson correlation coefficient will be used for correlation analysis; otherwise, the Spearman correlation coefficient will be used. Boxplots will be used to show the distribution of biomarker levels by cyst type, Scatter Plots will be used to visualize correlations between biomarkers, and Bar Graphs will be used to compare mean biomarker levels by cyst type.

The underlying mechanism of odontogenic tumors and cysts is not yet clear. In the literature review, no studies were found on MMP-8 in odontogenic tumors, and only a few studies were found on RANKL and MIP-1alpha. Therefore, the aim of this study is to gain insight into cyst pathology by examining the levels of biomarkers in odontogenic cyst fluid. The secondary objective of this study is to examine the correlation between markers measured by cyst type.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals diagnosed with cysts
2. Individuals who are not pregnant or breastfeeding
3. Individuals who agree to sign the informed consent form

Exclusion Criteria:

1. Systemically ill individuals who are contraindicated for surgery.
2. Individuals who do not wish to sign the informed consent form.
3. Individuals who are pregnant, breastfeeding, or using oral contraceptives will be excluded.

Ages: 12 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study group will consist of individuals aged 12-80 with cystic lesions who agree to participate in the study themselves and with their families (if children), and who are not pregnant or breastfeeding.
Sampling Method: Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2025-08-25 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
MMP-8 concentration level in cyst fluid | through study completion, an average of 6 months
  Cyst fluids aspirated during the puncture will be centrifuged using a centrifuge and stored at -80 degrees Celsius in Eppendorf tubes until examined. After all samples are collected, the MMP-8 concentration level will be measured.
MMP-9 concentration level in cyst fluid | through study completion, an average of 6 months
  Cyst fluids aspirated during the puncture will be centrifuged using a centrifuge and stored at -80 degrees Celsius in Eppendorf tubes until examined. After all samples are collected, the MMP-9 concentration level will be measured.
RANKL concentration level in cyst fluid | through study completion, an average of 6 months
  Cyst fluids aspirated during the puncture will be centrifuged using a centrifuge and stored at -80 degrees Celsius in Eppendorf tubes until examined. After all samples are collected, the RANKL concentration level will be measured.
MIP-1alpha concentration level in cyst fluid | through study completion, an average of 6 months
  Cyst fluids aspirated during the puncture will be centrifuged using a centrifuge and stored at -80 degrees Celsius in Eppendorf tubes until examined. After all samples are collected, the MIP-1alpha concentration level will be measured.

SECONDARY OUTCOMES:
Correlation between the type of cyst and the measured markers | through study completion, an average of 6 months
  After measuring the concentration levels of the MMP-8, MMP-9, RANKL, and MIP-1alpha biomarkers in the cyst fluid, the results will be compared with the subsequent biopsy results to examine their correlation with the type and origin of the cyst.

CONTACTS AND LOCATIONS:
Overall Officials: hande has elci, Principal Investigator — Harran University
Locations (1):
- Harran University, Faculty of Dentistry, Sanliurfa, Turkey (Türkiye)